CLINICAL TRIAL: NCT01858688
Title: A Phase II, Prospective Study of MRI in the Reclassification of Men Considering Active Surveillance in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Neil Martin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-056
Record Dates: First submitted 2013-05-15; First posted 2013-05-21 (Estimated); Results first posted 2022-05-18 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; MRI; Active surveillance in prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Evaluation of accuracy of the MRI relative to biopsy
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Accuracy of multi-parametric MRI relative to prostate biopsy (Experimental): Determine the sensitivity and specificity of MP-erMRI relative to repeat 12 core TRUS biopsy for classifying upgrading of disease extent or Gleason grade in men considering AS.
  Interventions: Device: Multiparametric MRI; Procedure: Prostate biopsy

INTERVENTIONS:
Device: Multiparametric MRI — an MRI of the prostate will be performed
Procedure: Prostate biopsy — a biopsy of the prostate will be performed according to standard procedures for men on active surveillance

SUMMARY:
Some men newly diagnosed with prostate cancer do not require immediate treatment. Rather, they can be followed closely with regular physical exams, blood work and repeated biopsies of the prostate. If the prostate cancer is becoming more aggressive, curative treatment can be offered at that time. This strategy of delaying treatment until necessary is called active surveillance in prostate cancer.

Active surveillance is a way of monitoring prostate cancer which aims to avoid or delay unnecessary treatment in men with less aggressive cancer.

Prostate cancer can be slow growing and, for many men, the disease may never progress or cause any symptoms. In other words, many men with prostate cancer will never need any treatment. Treatments for prostate cancer may cause side effects which can affect your quality of life. By monitoring the cancer with regular tests, you can avoid or delay these side effects.

Active surveillance is generally suitable for men with low risk early stage prostate cancer that is contained within the prostate gland (localized prostate cancer).

If doctors had a better way of identifying who might be best suited for this approach, it would likely become more appealing for more men. In this study, the investigators are looking at how accurate a magnetic resonance imaging (MRI) scan is at identifying high-risk prostate cancer, which might make a man a poor candidate for active surveillance.

To do this, the investigators are collecting data from the MRI scan of men and comparing it to a trans-rectal biopsy performed following the scan. The results of this study will help inform doctors how accurate the MRI is in identifying men who should not be on active surveillance.

DETAILED DESCRIPTION:
Before the research starts (screening): After signing this consent form, you will be asked to undergo some screening tests or procedures to find out if you can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated.

* A medical history, which includes questions about your health, current medications, any allergies and evaluation for whether you can safely have an MRI and biopsy
* Performance status, which evaluates how you are able to carry on with your usual activities.
* Review of the initial diagnostic biopsy, which you had when you were diagnosed with prostate cancer.
* Routine Blood Tests ( PSA is a protein that is produced by the prostate gland. The PSA test has been widely used to screen men for prostate cancer. It is also used to monitor men who have been diagnosed with prostate cancer to see if their cancer is responding to therapy)
* Physical Exam
* Health State Questionnaires
* These questionnaires review: Your feelings about your cancer diagnosis, your satisfaction with the cancer care you received, your health and symptoms over the past four weeks, and your overall urinary function

If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

After the screening procedures confirm that you are eligible to participate in the research study:

* You will be scheduled for a MRI between 2 to 14 months after your initial biopsy, which showed prostate cancer, to assess the grade and extent of your prostate cancer since your initial diagnosis.
* You will be scheduled for a repeat prostate biopsy 0-3 months after your MRI is reviewed.

Based on the findings from the MRI, this biopsy will be performed either in the urologist's office with an ultrasound (a medical imaging technique that uses high frequency sound waves and their echoes) or using anesthesia and an MRI to guide where the biopsy is taken within the prostate.

If the MRI does not show anything of concern, you will have another ultrasound-guided biopsy similar to the one you had when you were initially diagnosed with prostate cancer. In this procedure twelve biopsy samples are taken from the prostate. Each biopsy is about the length of a dime and as narrow as a toothpick.

If the MRI has findings which need further evaluation, you will have a guided biopsy. In this procedure, you will have twelve samples taken from the prostate similar to the biopsy you had when you were diagnosed with prostate cancer. Additionally, several biopsies will be taken of the area or areas of concern noted on the MRI. This procedure will require anesthesia, which may be general anesthesia or another type. You will meet with the study physician prior to the biopsy procedure. The type of anesthesia to be used will be decided by the study physician in discussion with you. When undergoing a study in the MRI system, you will lie motionless inside this device Occasionally the machine will produce a loud banging noise, as if it were being pounded from the outside with a hammer. Earplugs are available to reduce this sound level.

While you are in the magnet, under the anesthetic, the investigators will do the biopsy. To do this the investigators will use 2 ways to help us reach the correct part of your prostate, one is a robotic needle holder, which will show us where to put the needle, by lining up the correct place outside on the skin or rectal wall and the study physician will push in the needle with his/her hand. Second the investigators will use a model of the best location(s), taken from images. The biopsy is done with a needle put in through the skin, under your scrotum or through the rectal wall by the doctor.

The entire length of the procedure will be approximately 3 hours. The results of the procedure and biopsy will be communicated by your doctor as soon as they are available. The results will also be shared with the research co-investigators. This will be done by sharing the pathology results for each biopsy as matched with the location/place it came from in your gland. The study doctor will share the results of your biopsy with you at your end of study visit.

Medical Information The investigators will collect your medical information when you come to the Dana-Farber Cancer Institute and link this information to your specimens so that the investigators may better understand how these tests affect how participants do over time. It is important to note the following: all blood, tissue, and data collected from participants will be used for research only and when the research is performed on your samples, the investigators conducting this research will not have access to participant identification information, such as medical record numbers.

End of study visit:

You will have an end of study visit approximately 30 days after your final biopsy is performed. At this visit, the study staff will:

* Review your current PSA lab values
* Review the results of your biopsy and discuss options for future treatment.
* Ask you to complete several "Health- State" questionnaires if you have not already done so
* Review any side effects that you may have experienced as a result of your recent biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* The subject will have histologically confirmed prostate cancer with all of the following features:
* Minimum 10 core prostate biopsy showing histologically-confirmed prostate cancer within 12 months of enrollment reviewed by a pathologist from one of the DF/HCC associated hospitals
* Gleason ≤3+3
* No tertiary Gleason grade ≥4
* ≤3 total cores positive
* ≤50% of any given core involved with cancer
* No evidence on biopsy of extracapsular extension
* PSA within one month of enrollment: <10 ng/mL
* Clinical stage: ≤T2a & N0 or NX & M0
* The subject is able and willing to abide by the study protocol or cooperate fully with the investigator or designee
* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document
* Age ≥18
* Life expectancy of greater than 10 years
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* First diagnosis of prostate cancer > 12 months prior to enrollment
* Prior prostate cancer-directed therapy including:
* androgen deprivation therapy
* radiation therapy to the prostate (external beam or brachytherapy)
* cryotherapy
* high-intensity focused ultrasound (HIFU)
* chemotherapy for prostate cancer
* Prior transurethral resection of prostate
* Subject who is deemed by the treating physician to have a contraindication to definitive treatment
* Subjects with a contraindication to an MRI including those with a pacemaker, ferromagnetic aneurysm clip, or cochlear implants
* Subjects with a contraindication to receiving Gadolinium containing contrast for the MRI
* Conditions which make repeat TRUS biopsies not feasible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-09; Primary Completion 2018-05 (Actual); Study Completion 2023-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil E Martin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2013 - May 2017
Period: Overall Study
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
Started | 101
Biopsied at Baseline | 97
MRI Assessed | 91
Completed (Participants with TRUS biopsy at baseline as well as MRI and TRUS Biopsy post-baseline) | 81
Not Completed | 20
Not completed — Withdrawal by Subject | 8
Not completed — Participant began another therapy | 3
Not completed — Physician Decision | 2
Not completed — Progressive Disease | 2
Not completed — Reason not reproted | 5

BASELINE CHARACTERISTICS:
Population: Population with baseline data
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
Number analyzed (Participants) | 97
Age, Continuous [Median (Full Range); unit: years] | 58 [47 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 90
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 87
  More than one race | 0
  Unknown or Not Reported | 5
Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status was used
  Participants
    0 - Fully Active | 87
    1 - Restricted | 1
    Missing | 9
Prostate-Specific Antigen Titer [Median (Full Range); unit: ng/mL] | 4.6 [0.6 to 9.2]
Clinical Stage [Count of Participants; unit: Participants] — T1: Tumor not visible on imaging T1a: Cancer in <5% of cells removed during benign prostate hyperplasia (BPH) surgery T1b: Cancer in >5% of cells removed during BPH surgery. T1c: Tumor found during needle biopsy T2a: Tumor has invaded 1/2 or less of one side of the prostate T2b: Tumor has invaded more than 1/2 of one side of the prostate T2c: Tumor has invaded both sides of the prostate T3: Tumor has developed outside of the prostate and may have spread to the seminal vesicles T4: Tumor has spread beyond the seminal vesicle (rectum, bladder, urethral sphincter, pelvic wall)
  Participants
    T1a | 0
    T1b | 0
    T1c | 83
    T2a | 11
    T2b | 0
    T2c | 0
    T3 | 0
    T4 | 0
    Missing | 3
Adult Comorbidity Evaluation Index [Count of Participants; unit: Participants] — The score can be none (0), mild (1), moderate (2) or severe (3) and is defined according to the highest scored ailment. In cases with two or more grade 1 ailments, a final score of 1 assigned. In cases with two or more grade 2 ailments in different organ systems, a final score of 3 is assigned.
  Participants
    None | 23
    Mild | 30
    Moderate | 27
    Severe | 2
    Unknown | 15
Computerized Tomography (CT) of Abdomen and Pelvis [Count of Participants; unit: Participants]
  Yes | 6
  No | 91
CT Bone Scan [Count of Participants; unit: Participants]
  Yes | 3
  No | 94
Gleason Score [Count of Participants; unit: Participants] — The pathologist looking at the biopsy sample will assign one Gleason grade to the most predominant pattern in your biopsy and a second Gleason grade to the second most predominant pattern. For example: 3 + 4. The two grades will then be added together to determine your Gleason score. Theoretically, Gleason scores range from 2-10. However, since Dr. Gleason's original classification, pathologists almost never assign scores 2-5, and Gleason scores assigned will range from 6 to 10, with 6 being the lowest grade cancer.
  Participants
    3+3 | 97
    Missing | 0
Evidence of Perineural Invasion [Count of Participants; unit: Participants]
  Yes | 4
  No | 92
  Missing | 1
Extracapsular Extension [Count of Participants; unit: Participants]
  Yes | 0
  No | 93
  Missing | 4

OUTCOME MEASURES:

1. Primary Outcome: MP-erMRI Classification Sensitivity
Description: The classification sensitivity of multiparametric endorectal magnetic resonance imaging (MP-erMRI) when compared to the standard of care procedure (transrectal ultrasound-guided (TRUS) re-biopsy) The sensitivity is equivalent to the proportion of patients who were reclassified by MP- erMRI out of the total number of patients who should have been reclassified (given their TRUS re-biopsy result). In other words, it is the proportion of participants reclassified appropriately by MP- erMRI.
Time Frame: From baseline biopsy to final biopsy, up to 18 months
Population: Population that completed all treatment interventions.
Measure: Number (90% Confidence Interval); unit: proportion of true positives
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
Number analyzed (Participants) | 81
proportion of true positives | 0.875 [0.656 to 0.977]

2. Primary Outcome: MP- erMRI Classification Specificity
Description: The classification specificity of multiparametric endorectal magnetic resonance imaging (MP-erMRI) when compared to the standard of care procedure (transrectal ultrasound-guided (TRUS) re-biopsy) The specificity is equivalent to the proportion of patients who were not reclassified by MP- erMRI out of the total number of patients who should have been not reclassified (given their TRUS re-biopsy result). In other words, it is the proportion of participants not reclassified appropriately by MP- erMRI.
Time Frame: From baseline biopsy to final biopsy, up to 18 months
Population: Population that completed all treatment interventions.
Measure: Number (90% Confidence Interval); unit: proportion of true negatives
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
Number analyzed (Participants) | 81
proportion of true negatives | 0.785 [0.684 to 0.865]

3. Secondary Outcome: Frequency of Reclassification
Description: The frequency of reclassification using MP- erMRI, given in the form of a percentage of participants who have been reclassified.
Time Frame: From baseline biopsy to final MRI, up to 18 months
Population: The population that underwent MRI
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
Number analyzed (Participants) | 90
percentage of participants | 40 [31.3 to 49.2]

4. Secondary Outcome: Median Change in Illness-Related Uncertainty, Anxiety, and Distress
Description: The median change from baseline in illness-related uncertainty, anxiety, and distress measured by The Mishel Uncertainty in Illness Scale Community Form for Active Surveillance (MUIS-AS). The questionnaire entails 15 parts scored from 0-4 for a total of 0-60. The higher the score, the worse the symptoms of uncertainty, anxiety, and distress.
Time Frame: From baseline biopsy to final MRI, up to 18 months
Population: Baseline and post-study questionnaire data available for 48 participants.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
Number analyzed (Participants) | 48
score on a scale | -2 [-27 to 12]

5. Secondary Outcome: Median Change in Service Satisfaction
Description: The median change from baseline in service satisfaction measured by Services Satisfaction Scale - for Cancer Care (SSS-Ca). The questionnaire entails 5 parts scored from 1-7 for a total of 7-35. The higher the score, the more dissatisfied the participant.
Time Frame: From baseline biopsy to final MRI, up to 18 months
Population: Baseline and post-study questionnaire data available for 47 participants.
Measure: Median (Full Range); unit: change in score
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
Number analyzed (Participants) | 47
change in score | 0 [-9 to 19]

6. Secondary Outcome: Median Change in Prostate Cancer Symptoms
Description: The median change from baseline in prostate cancer symptoms measured by the Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP). The questionnaire entails 15 parts scored from 0-4 for a total of 0-60. The higher the score, the worse the symptoms.
Time Frame: From baseline biopsy to final MRI, up to 18 months
Population: Baseline and post-study questionnaire data available for 47 participants.
Measure: Median (Full Range); unit: change in score
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
Number analyzed (Participants) | 47
change in score | 0 [-6 to 9.8]

7. Secondary Outcome: Median Change in Urinary Symptoms
Description: The median change from baseline in urinary symptoms measured by the American Urological Association Symptoms Index (AUA SI). The questionnaire entails 8 parts. Parts 1-7 are scored 0-5 (for a total scoring range of 0-35) and part 8, a question evaluating psychological effect is scored from 0-6. The higher the score, the worse the participant's symptoms.
Time Frame: From baseline biopsy to final MRI, up to 18 months
Population: Baseline and post-study questionnaire data available for 49 participants. Only 46 participants have complete data for question 8.
Measure: Median (Full Range); unit: change in score
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
Number analyzed (Participants) | 49
change in score
  Urinary Symtoms | 0 [-7 to 10]
  Psychological Effect: number analyzed (Participants) | 46
  Psychological Effect | 0 [-2 to 2]

8. Secondary Outcome: Disease Extent by Classification Status
Description: Disease extent evaluated using established methods and given here by MP- erMRI classification status.
Time Frame: From baseline biopsy to final biopsy, up to 18 months
Population: All the available targeted biopsy results are 'Not Reclassified', without any input from the other category, no comparison can be made.
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
Number analyzed (Participants) | 0

9. Secondary Outcome: Gleason Score by Classification Status
Description: Gleason Score evaluated using established methods and given here by MP- erMRI classification status.
Time Frame: From baseline biopsy to final biopsy, up to 18 months
Population: as for outcome 8
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From biopsy to exit visit, up to 20 months.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. Remaining AEs are classified as Other AEs (OAE). Maximum grade toxicity by type was calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term. Participants are not being evaluated based on their post-operative treatment option.
Arm/Group | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy
All-Cause Mortality (participants affected / at risk) | 0/97
Serious Adverse Events (participants affected / at risk) | 2/97
Other Adverse Events (participants affected / at risk) | 4/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy (N=97)
Syncope (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 1
Prostate Infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Accuracy of Multi-parametric MRI Relative to Prostate Biopsy (N=97)
Hematuria (Renal and urinary disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT01858688/Prot_SAP_000.pdf